CLINICAL TRIAL: NCT05048004
Title: Cerebral Embolization During Pulmonary Vein Isolation: an Observational Study
Brief Title: Cerebral Embolization During Pulmonary Vein Isolation
Acronym: TCD-CA
Status: Recruiting | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Christian Nolte, Principal Investigator, Charite University, Berlin, Germany
Other Study IDs: EA1/215/20
Record Dates: First submitted 2021-08-09; First posted 2021-09-17 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Atrial Fibrillation; Ischemic Stroke; Cerebral Microembolism
MeSH Terms: conditions — Atrial Fibrillation; Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- QMODE intervention: catheter ablation performed using high-power with a maximum of up to 50 W (QMODE) and
  Interventions: Procedure: QMODE intervention
- QMODE+ intervention: catheter ablation performed using very high power with a maximum of up tp 90 W (QMODE +)
  Interventions: Procedure: QMODE+ intervention

INTERVENTIONS:
Procedure: QMODE intervention — Patients undergoing different forms of pulmonary vein isolation are being monitored for microembolic signals (MES) by transcranial ultrasound. For standard ablation, a Thermocool Smarttouch SF (Biosense Webster) catheter will be used (50 W, target ablation index of 550).
  Groups: QMODE intervention
Procedure: QMODE+ intervention — Patients undergoing different forms of pulmonary vein isolation are being monitored for microembolic signals (MES) by transcranial ultrasound. For comparison, catheter ablation performed using very high power with a maximum of up tp 90 W (QMODE +) will be used.
  Groups: QMODE+ intervention

SUMMARY:
The goal of the TCD-CA study is to determine the frequency of cerebral embolization during pulmonary vein isolation using continuous transcranial Doppler examination. Different parts of the procedure, different ablation techniques and periprocedural anticoagulation regimes will be compared.

DETAILED DESCRIPTION:
Pulmonary vein isolation (PVI) is a well-established interventional treatment of patients with atrial fibrillation. Previous studies have shown that catheter-based treatments such as PVI may lead to cerebral ischemia. Cerebral ischemia related to PVI may present with new neurological deficits but may also occur as "silent brain infarction". However, even "silent brain infarctions" are associated with an increased risk of incident dementia and clinically overt new strokes. To date, it remains unclear which procedural steps of PVI are associated with an increased risk of cerebral ischemia.

Cerebral blood flow and microembolic signals can be detected by using transcranial doppler ultrasound (TCD). TCD has been used in clinical routine for many years and is known to be safe in stroke patients. By performing continuous TCD monitoring for microembolic signals during PVI, the aim of this study is therefore to identify, which procedural steps are associated with the occurence of cerebral microemboli. In addition, the investigators aim to compare the frequency of cerebral microemboli in different pulmonary vein isolation techniques, namely high-power with a maximum of up to 50 W (QMODE) and very high power with a maximum of up tp 90 W (QMODE +)

ELIGIBILITY:
Inclusion Criteria:

* patients with atrial fibrillation undergoing first-ever catheter-based ablation at Charité-Campus Benjamin Franklin
* age 18 years or older

Exclusion Criteria:

* pregnancy
* patient unable to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients who undergo pulmonary vein isolation as part of their treatment for atrial fibrillation at Charité-Campus Benjamin Franklin are eligible for study participation. Clinical indication for the procedure will be established by the treating physician prior to and irrespective of study participation. Patients who are unable to provide written informed consent will not be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Microembolic Signals (MES) | during the procedure
  number of MES detected by transcranial doppler ultrasound

SECONDARY OUTCOMES:
neurological outcome | at baseline, 0-5 days after pulmonary vein isolation
  neurological outcome will be evaluated using the National Institute of Health Stroke Scale
cognitive outcome | at baseline, 0-5 days after pulmonary vein isolation
  cognitive outcome will be evaluated using the Montreal Cognitive Assessment
cerebral infarctions | at baseline, 0-5 days after pulmonary vein isolation
  number of new cerebral infarctions on magnetic resonance imaging
cerebral microbleeds | at baseline, 0-5 days after pulmonary vein isolation
  number of new cerebral microbleeds on magnetic resonance imaging
cerebral macrobleeds | at baseline, 0-5 days after pulmonary vein isolation
  number of new cerebral macrobleeds on magnetic resonance imaging

CONTACTS AND LOCATIONS:
Overall Officials: Christian H Nolte, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité-University Medicine Berlin, Campus Benjamin Franklin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No